CLINICAL TRIAL: NCT03074955
Title: Preventive Effect of Leg Wrapping Combined With Trendelenburg Position on Hypotension Induced by Propofol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyungmook Lee (Other)
Responsible Party: Sponsor-Investigator, Hyungmook Lee, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1304200001
Record Dates: First submitted 2017-02-26; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Hypotension; Propofol
Keywords: Hypotension; Propofol; Trendelenburg; leg wrapping
MeSH Terms: conditions — Hypotension | interventions — Head-Down Tilt; Supine Position

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): leg wrapping without tension & maintain supine position
  1. Apply elastic bandages to both legs without tension.
  2. Maintain supine position after injecting propofol.
  3. After 3 minutes from propofol injection, remove elastic bandages
  4. induction using propofol 2mg/kg
  5. After bispectral index (BIS) goes below 60 & patient become unconsciousness, inject rocuronium 0.6mg/kg
  6. intubate patient between 3 and 4 minutes after propofol injection
  7. measure blood pressure ( systolic, diastolic, mean ) & heart rate at 1,2,3,4,5 minutes after propofol injection
  8. phenylephrine injection if hypotension develops
  Interventions: Device: leg wrapping without tension; Procedure: supine position
- Trendelenburg only (Experimental): leg wrapping without tension & apply Trendelenburg position
  1. Apply elastic bandages to both legs without tension.
  2. After injecting propofol, apply Trendelenburg position ( 10 degree )
  3. After 3 minutes from propofol injection, remove elastic bandage and revert to supine position.
  4. induction using propofol 2mg/kg
  5. After bispectral index (BIS) goes below 60 & patient become unconsciousness, inject rocuronium 0.6mg/kg
  6. intubate patient between 3 and 4 minutes after propofol injection
  7. measure blood pressure ( systolic, diastolic, mean ) & heart rate at 1,2,3,4,5 minutes after propofol injection
  8. phenylephrine injection if hypotension develops
  Interventions: Procedure: Trendelenburg position; Procedure: supine position
- Trendelenburg & leg wrapping (Experimental): leg wrapping with tension & apply Trendelenburg position
  1. Apply elastic bandages to both legs with tension.
  2. After injecting propofol, apply Trendelenburg position ( 10 degree )
  3. After 3 minutes from propofol injection, remove elastic bandage and revert to supine position.
  4. induction using propofol 2mg/kg
  5. After bispectral index (BIS) goes below 60 & patient become unconsciousness, inject rocuronium 0.6mg/kg
  6. intubate patient between 3 and 4 minutes after propofol injection
  7. measure blood pressure ( systolic, diastolic, mean ) & heart rate at 1,2,3,4,5 minutes after propofol injection
  8. phenylephrine injection if hypotension develops
  Interventions: Device: leg wrapping with tension; Procedure: Trendelenburg position

INTERVENTIONS:
Device: leg wrapping with tension — 1. Apply elastic bandages with tension to both legs before injecting propofol.
  2. After 3 minutes, remove elastic bandages.
  Arms: Trendelenburg & leg wrapping
Procedure: Trendelenburg position — 1. Apply Trendelenburg position positon of 10 degree after injectin propofol
  2. After 3 minutes, change to supine position
  Arms: Trendelenburg & leg wrapping; Trendelenburg only
Device: leg wrapping without tension — 1. Apply elastic bandages without tension to both legs before injecting propofol.
  2. After 3 minutes, remove elastic bandages
  Arms: Control
Procedure: supine position — 1.maintain supine position
  Arms: Control; Trendelenburg only

SUMMARY:
Although propofol is widely used as an induction agent for a general anesthesia, it can induce a profound hypotension, which leads to the hypo-perfusion of end organs and eventually increases morbidities. Theoretically, applying Trendelenburg position (head down and leg up position) increases cardiac preloads and cardiac outputs. However, in past researches, changing to Trendelenburg position alone is not enough and does not prevent propofol induced hypotension. Previous studies proved that leg wrapping effectively prevent hypotension after neuraxial anesthesia during Cesarean section. The leg wrapping prevents hypotension by increasing vascular resistance of lower extremities. The investigators made a hypothesis that applying both Trendelenburg position and leg wrapping prevent propofol induced hypotension more effectively than either applying Trendelenburg position only or taking no preventive measures.

DETAILED DESCRIPTION:
** Study procedure

1. check baseline blood pressure ( systolic, diastolic, mean) and heart rate.
2. apply pre-defined measures to each group(arm) ( summarized in arms and interventions section )
3. induction using propofol 2mg/kg
4. After bispectral index (BIS) goes below 60 & patient become unconsciousness, inject rocuronium 0.6mg/kg
5. intubate patient between 3 and 4 minutes after propofol injection
6. measure blood pressure ( systolic, diastolic, mean ) & heart rate at 1,2,3,4,5 minutes after propofol injection
7. phenylephrine injection if hypotension develops

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic status class 1, 2, and 3.
* under general anesthesia

Exclusion Criteria:

* severe cardiac/pulmonary/liver/renal disease
* BMI > 30 kg/m2
* known or risk factor of increased intraocular pressure or intracranial pressure
* uncontrolled hypertension
* high risk for propofol allergy
* allergies to medications related to anesthesia
* mechanical difficulties with leg wrapping ( wound on legs, devices on legs )
* emergent operation
* high risk of gastric aspiration ( gastrointestinal obstruction, short nil per os(NPO) time )
* patient wearing elastic stocking for therapeutic purpose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2013-08-16 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
SBP_2 | 2 minutes from propofol injection
  systolic blood pressure at 2 minutes from propofol injection

CONTACTS AND LOCATIONS:
Overall Officials: MiHyun Kim, Dr. PhD., Study Director — Department of anesthesia and pain medicine, Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seo-Cho Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun HL, Ling QD, Sun WZ, Wu RS, Wu TJ, Wang SC, Chien CC. Lower limb wrapping prevents hypotension, but not hypothermia or shivering, after the introduction of epidural anesthesia for cesarean delivery. Anesth Analg. 2004 Jul;99(1):241-245. doi: 10.1213/01.ANE.0000121346.33443.5A. PMID 15281537
- [Background] Reuter DA, Felbinger TW, Schmidt C, Moerstedt K, Kilger E, Lamm P, Goetz AE. Trendelenburg positioning after cardiac surgery: effects on intrathoracic blood volume index and cardiac performance. Eur J Anaesthesiol. 2003 Jan;20(1):17-20. doi: 10.1017/s0265021503000036. PMID 12553383